CLINICAL TRIAL: NCT01981174
Title: The Effect of Needle Size on Pain Perception in Patients Treated With Botulinum Toxin A Injections
Brief Title: A Pilot Study of Needle Size and Pain Perception With Botulinum Toxin A Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: STU84470
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30-gauge needle (Active Comparator): Subjects will be screened, assessed, and randomized to be injected with onabotulinum toxin A using a 30-gauge needle on one side of the face and injected using a 32-gauge needle on the other side during their first clinic visit. All needles would be luer lock, ½ inch length, and attached to separate 1cc syringes. Injection depth would be 1-2mm, dermal, and the angle of incidence would be perpendicular.
  Interventions: Procedure: 30-gauge needle
- 32-gauge needle (Active Comparator): Subjects will be screened, assessed, and randomized to be injected with onabotulinum toxin A using a 30-gauge needle on one side of the face and injected using a 32-gauge needle on the other side during their first clinic visit. All needles would be luer lock, ½ inch length, and attached to separate 1cc syringes. Injection depth would be 1-2mm, dermal, and the angle of incidence would be perpendicular.
  Interventions: Procedure: 32-gauge needle

INTERVENTIONS:
Procedure: 30-gauge needle
  Arms: 30-gauge needle
Procedure: 32-gauge needle
  Arms: 32-gauge needle

SUMMARY:
The purpose of this study is to compare the levels of pain resulting from injections of Botox® for wrinkles on the forehead and between the eyes using two different sized needles (32 gauge and 30 gauge needles).

DETAILED DESCRIPTION:
Subjects will be screened, assessed, and randomized to be injected with onabotulinum toxin A using a 30-gauge needle on one side of the face and injected using a 32-gauge needle on the other side during their first clinic visit. This study is a pilot study designed to determine feasibility of these procedures.

ELIGIBILITY:
Inclusion Criteria:

1. In good health
2. Is a female
3. Is 25-70 years of age
4. Has moderate dynamic forehead/glabellar wrinkles
5. Has willingness and the ability to understand and provide informed consent and communicate with the study staff

Exclusion Criteria:

1. Younger than 25 or older than 70 years of age
2. Pregnant or lactating
3. Is a male
4. Has received the following treatments in the forehead or glabellar region:

   1. botulinum toxin injections in the past 6 months
   2. ablative laser procedure in the past 6 months
   3. radiofrequency device treatment in the past 6 months
   4. ultrasound device treatment in the past 6 months
   5. medium to deep chemical peel in the past 6 months
   6. temporary soft tissue augmentation material in the area to be treated in the past year
   7. semi-permanent soft tissue augmentation material in the area to be treated in the past 2 years
   8. permanent soft tissue augmentation material in the area to be treated
5. Has an active infection in the forehead or glabellar region (excluding mild acne)
6. Is allergic to cow's-milk protein
7. Is allergic to albumin
8. Taking aminoglycoside
9. Is currently using anticoagulation therapy
10. Has a history of bleeding disorders
11. Has a mental illness
12. Unable to understand the protocol or to give informed consent

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Visual analog score (VAS) pain rating after each side is injected | 1 hour on Treatment day
  Subjects will rate pain using the visual analog score (VAS 1-10) after each side is injected using the 30 or 32 gauge needles. Lower values represents less pain; higher values represents more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Derived] Alam M, Geisler A, Sadhwani D, Goyal A, Poon E, Nodzenski M, Schaeffer MR, Tung R, Minkis K. Effect of Needle Size on Pain Perception in Patients Treated With Botulinum Toxin Type A Injections: A Randomized Clinical Trial. JAMA Dermatol. 2015 Nov;151(11):1194-9. doi: 10.1001/jamadermatol.2015.2232. PMID 26352252